CLINICAL TRIAL: NCT04833751
Title: Registry of Cardiovascular Anesthesia Including the Database of Biological Signals During Anesthesia, Preoperative Assessment and Prognosis in Patients: Severance Cardiovascular Surgery Prospective (SECURE) Database
Brief Title: Registry of Cardio/Neurovascular Anesthesia Including the Database of Biological Signals During Anesthesia, Preoperative Assessment and Prognosis in Patients
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-1002
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Anaesthesia
Keywords: Cardiac Diseases; Biosignal data; Cardiac Surgical Procedures; Cardiovascular Surgical Procedures; Heart Valve Prosthesis Implantation
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anesthesia for cardiovascular surgery or procedure: Patients undergoing anesthesia in an operating room or hybrid room for cardiovascular surgery or procedure.

SUMMARY:
The purpose of this study is to establish a registry database for patients undergoing anesthesia for cardiovascular surgery or procedures in our operating or hybrid room. The following information will be collected:

1. Preoperative patient assessment
2. All monitored perioperative biosignal data
3. Intraoperative and immediate postoperative hemodynamic information, input/output balance, and medication usage
4. Short- and long-term prognosis from electronic medical records This database will be used to develop a vigilant monitoring system that integrates multiple biosignal data simultaneously, contributing to the improvement of anesthesia care.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 19 and older
2. Patients scheduled for anesthesia at a cardiovascular hospital for cardiovascular surgery or procedures

Exclusion Criteria:

1) Emergency (surgery/procedure room transfer within 1 hour of visit) where there is insufficient time for the subject (adult 19 years of age or older) or his/her representative (adult incapable of consent) to decide whether to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardio/neurovascular surgery or procedure
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year after surgery
  All-cause mortality within one year after surgery

SECONDARY OUTCOMES:
Postprocedural myocardial infarction | within 2days after surgery
  Defined by an increase in CK-MB or cardiac troponin (cTn) levels.
Acute kidney injury | within 7days after surgery
  The definition of AKI refers to the Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group's KDIGO Clinical Practice Guideline for Acute Kidney Injury.
surgical re-exploration | within 30 days (±3 days) after surgery
  require a return to the operating room for bleeding with or without tamponade, graft occlusion, valve dysfunction, or other cardiac reason
deep sternal wound infection | within 30 days (±3 days) after surgery
  infection involving muscle, bone, or mediastinum requiring operative intervention
prolonged mechanical ventilation | within 30 days (±3 days) after surgery
  intubation required for more than 24 hours
stroke/cerebrovascular accident | within 30 days (±3 days) after surgery
  Confirmed neurological deficit caused by a blood supply disturbance to the brain lasting more than 24 hours
Readmission rate | within 30days of the date of discharge from the index cardiac surgery hospitalization
  readmission to an acute care hospital within 30 days of discharge from the cardiac surgery hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Soh, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
  Start and end dates: Beginning 6 months and ending 36 months following article publication.